CLINICAL TRIAL: NCT04309344
Title: Biological Effects of a Bipolar Radiofrequency-based Device Over Shoulder Cartilage - a Randomized Controlled Clinical Trial
Brief Title: Biological Effects of a Bipolar Radiofrequency-based Device Over Shoulder Cartilage
Acronym: Alexsen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 831
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Glenohumeral Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RF (Experimental): The bipolar radiofrequency-based chondroplasty device is used in the COBLATION mode (yellow) with The WEREWOLF system and the wand FLOW 50 in Lo mode (low) which are approved by the FDA for chondroplasty and debridement of the articular cartilage
  Interventions: Device: WEREWOLF COBLATION System
- Control (Active Comparator): The mechanical shaver is used to remove superficial fibrillations.
  Interventions: Procedure: control

INTERVENTIONS:
Device: WEREWOLF COBLATION System — The bipolar radiofrequency-based chondroplasty device is used in the COBLATION mode (yellow) with The WEREWOLF system and the wand FLOW 50 in Lo mode (low) which are approved by the FDA for chondroplasty and debridement of the articular cartilage; fibrillations were removed and the surface was smoothed. This low energy and low suction setting minimizes damage to healthy chondrocytes surrounding and is therefore the preferred setting for the removal of articular cartilage.
  Arms: RF
Procedure: control — mechanical debridement
  Arms: Control

SUMMARY:
In the non-weight bearing glenohumeral joint, focal chondral defects are encountered infrequently and are usually found in association with other pathologies, such as glenohumeral instability, postoperative chondrolysis, focal osteonecrosis, septic arthritis, osteochondritis dissecans, and rotator cuff tears. Several studies revealed that approximately one-third of patients with rotator cuff disease have concomitant articular cartilage lesions. Because the glenohumeral articular cartilage is one of the thinnest in the body, the overall accuracy of non-contrast MRI in detecting glenohumeral articular cartilage lesions is moderate and it is difficult to have an accurate characterization of a lesion my MRI. So, currently, arthroscopy is considered the ''gold standard'' for glenohumeral cartilage assessment. Even if the literature lacks high-quality evidence regarding the nonsurgical and surgical treatment options for patients with shoulder chondral defects, in these scenarios, where, in our experience, the most of the lesions are small, diffuse and of ICRS grade 2 or 3 (non-full thickness), arthroscopic debridement is a good option for addressing glenohumeral chondropathy. The main drawbacks with this type of procedure are the removal of underlying healthy cartilage and the potential lack of chondral surface smoothing. Alternatives used to perform arthroscopic chondral debridement is thermal application, carried out by the use of laser devices or the application of monopolar or bipolar radiofrequency (RF). As regards the glenohumeral joint, there are several studies that underlined the potential benefit of arthroscopic debridement in glenohumeral chondropathy and early stage of osteoarthritis, but the type of debridement used in all these studies was mechanical or not specified. Because recent studies showed that Compared to conventional MD, 50° RF treatment appears to be a superior method based on short- and medium-term clinical outcomes and the progression of knee osteoarthritis [11], we want to specifically evaluate the effects of RF in patients with grade II or III chondropathy found during arthroscopy for rotator cuff disorders.

DETAILED DESCRIPTION:
This study is a prospective, therapeutic open blind randomized study. The enrollment of the patients will start immediately after the ethical committee approval. Considering our cases and our experience we plan to reach 40 patients (20 patients for group) which respect the inclusion and exclusion criteria in 2 months. We plan to enroll 6 more patients (3 for each group) in order to cover eventual loss of patients during the follow-up and these patients will be evaluated after surgery only if there will not be any losses among the initial 40 patients. During surgery, assessment of the chondropathy will be done and only patients with International Cartilage Regeneration and Joint Preservation Society (ICRS) grade 2 or 3 chondropathy will be enrolled. After addressing the rotator cuff pathology, the patient will be randomized and the radio-frequency (RF) debridement will be performed or not performed, so the patients will enter the control group (no RF) or the treatment group. The clinical evaluation will be performed by R.R., preoperatively and at 3 months, 6 months and 12 months after surgery. At 3 months post-operatively an MRI will be obtained and assessed by an expert shoulder doctor with particular attention for the cartilage. All the data will be completed and analyzed in about 12-13 months after the enrollment is completed and we estimate to present the data by May 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50-70 years.
2. Arthroscopic surgery for rotator cuff disorders.
3. Arthroscopic findings of ICRS grade 2 or 3 chondropathy.
4. Ability to give informed consent according to the International Conference of Harmonization (ICH)-Good Clinical Practices (GCP), and national/local regulations.

Exclusion Criteria:

1. Patients with a diagnosis of osteoarthritis before surgery.
2. Patients with ICRS grade 4 chondropathy.
3. Patients who received subacromial decompression.
4. Patients who received biceps tenodesis after tenotomy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of pain reduction | 12 months after surgery
  it will be assessed with numeric rating scale (NRS) questionnaire (0 no ain-10 thw worst pain).

SECONDARY OUTCOMES:
Improvement of range of motion (ROM) | 12 months after surgery
  It will be evaluated during clinical examination using a goniometer in terms of forward flexion, abduction, external rotation with elbow at side (ER1), external rotation with elbow at 90° degree of abduction (ER2), and internal rotation (level reached from the hand on the back side)
Improvement of the subjective evaluation of the shoulder condition with the simple shoulder test (SST) | 12 months after surgery
  SST is a self-reported shoulder-specific questionnaire that measures functional limitations of the affected shoulder in patients with shoulder dysfunction. The SST consists of 12 questions with dichotomous (yes/ no) response options.
Improvement of the subjective evaluation of the shoulder condition and the pain with the Constant-Murley (CM) test | 12 months after surgery
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient (100 best shoulder condition-0 worst shoulder condition).
Improvement of the shoulder condition with the magnetic resonance imaging (MRI) | 3 months after surgery
  High resolution MRI will be acquired and evaluated by the radiologist

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Castagna, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No